CLINICAL TRIAL: NCT02066870
Title: Phase I Study of the Combination of Icotinib and Arsenic Trioxide in Treating Non-small-cell Lung Cancer Patients With Resistance to EGFR-TKI
Brief Title: Icotinib and Arsenic Trioxide in Treating Non-small-cell Lung Cancer Patients With Resistance to EGFR-TKI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV55
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Icotinib; Arsenic Trioxide; Resistance; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Arsenic Trioxide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib and arsenic trioxide (Experimental): Icotinib is administered 125 mg three times per day, until disease progression or untolerated toxicity.
  Arsenic trioxide is administered by intravenous injection with an initial dose of 4mg/m2 per day for day 1 to day 14 every 21 days.
  Three dose levels, 4mg/m2, 6mg/m2 and 8mg/m2 will be evaluated according to predefined dose escalation decision rules. The Maximum Administered Dose (MAD) was reached at the dose level when at least 2 patients developed a DLT. There was no further dose escalation when this dose was achieved.
  Interventions: Drug: Icotinib; Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Icotinib — Icotinib is administered orally 125 mg three times per day, until disease progression or untolerated toxicity.
  Other Names: BPI-9000; Commana
Drug: Arsenic trioxide — Arsenic trioxide is administered by intravenous injection with an initial dose of 4mg/m2 per day for day 1 to day 14 every 21 days.
  Three dose levels, 4mg/m2, 6mg/m2 and 8mg/m2 will be evaluated according to predefined dose escalation decision rules. The Maximum Administered Dose (MAD) was reached at the dose level when at least 2 patients developed a DLT. There was no further dose escalation when this dose was achieved.
  Other Names: Arsenic trioxide for injection

SUMMARY:
The NSCLC patients who experienced good clinical responses to an EGFR-TKI will inevitably develop acquired resistance. A great deal of research are focusing on this issue. Arsenic trioxide showed efficacy and safety in acute promyelocytic leukemia, multiple myeloma and other solid tumors. Moreover, preclinical studies showed arsenic trioxide can reduce the resistance of tumor cells to chemotherapy and TKIs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV lung cancer with EGFR mutation
* Progressed after platinum-based chemotherapy
* The last anti-tumor therapy before entering this study must be gefitinib, erlotinib or icotinib, and the duration for tumor response must be no less than 4 months, or the duration for stable disease must be no less than 6 months
* With a measurable disease with conventional CT) according to RECIST Criteria
* WHO performance status(PS)<= 2
* N>=1.5×109/L, Plt>=1.0×109/L,Hb>=9g/dL; AST&ALT should <2.5ULN(without liver metastasis) or <5ULN(with liver metastasis).TBIL<=1.5ULN.
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Allergic to icotinib or arsenic trioxide.
* Patients with metastatic brain tumors with symptoms.
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 8 weeks

SECONDARY OUTCOMES:
Progression-free survival | Up to 4 months
Time to death | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Saijuan Chen, MD, Principal Investigator — Ruijin Hospital; Yuankai Shi, MD, Principal Investigator — Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China